CLINICAL TRIAL: NCT04599296
Title: A Randomized Controlled Pilot Trial of Postoperative Hip Bracing After Arthroscopic Osteoplasty and Labral Repair for Femoroacetabular Impingement Syndrome
Brief Title: Postoperative Hip Bracing After Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Mia Hagen, Associate Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00010038; 5P30AR072572-02 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-22 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Femoroacetabular Impingement Syndrome; Acetabular Labral Tear
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Intervention Model Description: Patients randomized to wearing a hip brace after surgery 36 Patients randomized to not wearing a hip brace after surgery 36
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The treating surgeon, who is also the PI, will be blind to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hip Brace (Active Comparator): This group will be assigned to wear a hip brace post surgery.
  Interventions: Device: Hip brace
- No Intervention (No Intervention): This group will not be assigned a hip brace after surgery.

INTERVENTIONS:
Device: Hip brace — Hip brace
  Arms: Hip Brace

SUMMARY:
Hip arthroscopy for treatment of femoroacetabular impingement syndrome (FAIS) involves reshaping of the osseous sources of impingement ("osteoplasty") and treatment of impingement-associated labral tears with labral repair. Postoperative hip braces are advocated to decrease postoperative pain by offloading hip musculature. However there are no studies looking at efficacy of hip braces after hip arthroscopy, and on average 50% of high-volume hip arthroscopists use bracing. The objective of this study is to use a randomized controlled trial to test the cited benefits of postoperative hip bracing on short term patient reported pain scores, validated hip-specific pain scores, and physical exam findings of hip flexor tendonitis.

DETAILED DESCRIPTION:
Hip arthroscopy for treatment of femoroacetabular impingement syndrome (FAIS) involves reshaping of the osseous sources of impingement ("osteoplasty") and treatment of impingement-associated labral tears with labral repair. The hip joint is subluxated with traction to accomplish this procedure. The diagnoses of FAIS and the incidence of hip arthroscopy have both increased dramatically in the last 20 years in the US -- in a recent study using IBM Marketscan to evaluate rates of hip arthroscopic treatment of FAIS, the investigators found this incidence doubled from 1.2 to 2.1 per 100,000 person-years in just a 3-year period. Despite the increasing incidence of hip arthroscopy in the US, on a recent review the investigators have found few evidence-based studies on postoperative care. A particular area of debate is the use of postoperative hip braces. Postoperative hip braces are advocated to decrease postoperative pain by offloading hip musculature. They may also prevent overuse of the hip flexors by supporting the hip during gait. However there are no studies looking at efficacy of hip braces after hip arthroscopy, and on average 50% of high-volume hip arthroscopists use bracing. The utility of bracing is important because hip braces are expensive (averaging $350-$600): if there are over 7000 hip arthroscopies performed nationwide and 50% of surgeons use hip braces, this amounts to over $2,000,000. The investigator's overall objective is to use a randomized controlled trial to test the cited benefits of postoperative hip bracing on short term patient reported pain scores, validated hip-specific pain scores, and physical exam findings of hip flexor tendonitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 14-60 on date of surgery
* Patient seen at the institution for the study
* Patient scheduled to undergo arthroscopic osteoplasty and labral repair for femoroacetabular impingement syndrome.

Exclusion Criteria:

* Any patient anyone who cannot follow up in person in clinic for the 6-week postoperative visit.
* Non-English speaking patients (due to limited validation of the patient reported outcome measures in non-English speaking populations).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mia Hagen, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adib F, Johnson AJ, Hennrikus WL, Nasreddine A, Kocher M, Yen YM. Iliopsoas tendonitis after hip arthroscopy: prevalence, risk factors and treatment algorithm. J Hip Preserv Surg. 2018 Dec 24;5(4):362-369. doi: 10.1093/jhps/hny049. eCollection 2018 Dec. PMID 30647926
- [Background] Schairer WW, Nwachukwu BU, McCormick F, Lyman S, Mayman D. Use of Hip Arthroscopy and Risk of Conversion to Total Hip Arthroplasty: A Population-Based Analysis. Arthroscopy. 2016 Apr;32(4):587-93. doi: 10.1016/j.arthro.2015.10.002. Epub 2015 Dec 6. PMID 26671201
- [Background] Bozic KJ, Chan V, Valone FH 3rd, Feeley BT, Vail TP. Trends in hip arthroscopy utilization in the United States. J Arthroplasty. 2013 Sep;28(8 Suppl):140-3. doi: 10.1016/j.arth.2013.02.039. Epub 2013 Aug 1. PMID 23916639
- [Background] Yao JJ, Cook SB, Gee AO, Kweon CY, Hagen MS. What Is the Survivorship After Hip Arthroscopy for Femoroacetabular Impingement? A Large-database Study. Clin Orthop Relat Res. 2020 Oct;478(10):2266-2273. doi: 10.1097/CORR.0000000000001370. PMID 32604156
- [Background] Shin JJ, McCrum CL, Mauro CS, Vyas D. Pain Management After Hip Arthroscopy: Systematic Review of Randomized Controlled Trials and Cohort Studies. Am J Sports Med. 2018 Nov;46(13):3288-3298. doi: 10.1177/0363546517734518. Epub 2017 Oct 13. PMID 29028436
- [Background] Philippon MJ, Decker MJ, Giphart JE, Torry MR, Wahoff MS, LaPrade RF. Rehabilitation exercise progression for the gluteus medius muscle with consideration for iliopsoas tendinitis: an in vivo electromyography study. Am J Sports Med. 2011 Aug;39(8):1777-85. doi: 10.1177/0363546511406848. Epub 2011 May 12. PMID 21566069
- [Background] Domb BG, Sgroi TA, VanDevender JC. Physical Therapy Protocol After Hip Arthroscopy: Clinical Guidelines Supported by 2-Year Outcomes. Sports Health. 2016 Jul;8(4):347-54. doi: 10.1177/1941738116647920. Epub 2016 May 12. PMID 27173983
- [Background] Gupta A, Suarez-Ahedo C, Redmond JM, Gerhardt MB, Hanypsiak B, Stake CE, Finch NA, Domb BG. Best Practices During Hip Arthroscopy: Aggregate Recommendations of High-Volume Surgeons. Arthroscopy. 2015 Sep;31(9):1722-7. doi: 10.1016/j.arthro.2015.03.023. Epub 2015 May 14. PMID 25980403
- [Background] Cvetanovich GL, Lizzio V, Meta F, Chan D, Zaltz I, Nho SJ, Makhni EC. Variability and Comprehensiveness of North American Online Available Physical Therapy Protocols Following Hip Arthroscopy for Femoroacetabular Impingement and Labral Repair. Arthroscopy. 2017 Nov;33(11):1998-2005. doi: 10.1016/j.arthro.2017.06.045. Epub 2017 Sep 29. PMID 28969949
- [Background] Bolia IK, Briggs KK, Matheny L, Philippon MJ. Survey results from an international hip course: comparison between experts and non-experts on hip arthroscopy clinical practice and post-operative rehabilitation. Knee Surg Sports Traumatol Arthrosc. 2020 Apr;28(4):1270-1275. doi: 10.1007/s00167-018-5289-4. Epub 2018 Nov 22. PMID 30467580
- [Background] Truntzer JN, Shapiro LM, Hoppe DJ, Abrams GD, Safran MR. Hip arthroscopy in the United States: an update following coding changes in 2011. J Hip Preserv Surg. 2017 Mar 23;4(3):250-257. doi: 10.1093/jhps/hnx004. eCollection 2017 Aug. PMID 28948037
- [Background] Hagen M, Westermann R, Lynch T, Rosneck J. Rehabilitation for Femoroacetabular Impingement: Conservative Care and Postoperative Practice. J Hip Surg. 2018;02(04):189-193. doi:10.1055/s-0038-1676448
- [Derived] Hagen MS, Meier E, Wigton C, Son M, Kweon CY. A Randomized Controlled Trial of Postoperative Hip Bracing After Arthroscopic Osteoplasty and Labral Repair for Femoroacetabular Impingement Syndrome. Am J Sports Med. 2025 Dec;53(14):3332-3340. doi: 10.1177/03635465251388408. Epub 2025 Oct 30. PMID 41164948

RESULTS

PARTICIPANT FLOW:
Groups:
- No Brace: This group will not be assigned a hip brace after surgery.
Period: Overall Study
Arm/Group | Hip Brace | No Brace
Started | 41 | 41
Primary End Point (6 week postoperative) | 37 | 36
Completed (6 month postoperative) | 30 | 27
Not Completed | 11 | 14

BASELINE CHARACTERISTICS:
Population: Total number that reached postoperative at two weeks that had baseline data collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Hip Brace | No Intervention | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32 (10) | 34 (9) | 32.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] | 24 (5) | 27 (8) | 25.3 (7.0)
Smoking Status [Count of Participants; unit: Participants]
  Never | 27 | 29 | 56
  Quit | 9 | 8 | 17
  Current | 1 | 0 | 1
Marijuana Use [Count of Participants; unit: Participants]
  Never | 19 | 23 | 42
  Quit | 13 | 7 | 20
  Current | 5 | 7 | 12
Current Opioid Use [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 1
  No | 36 | 37 | 73
Duration of Symptoms [Count of Participants; unit: Participants]
  Less than 1 year | 10 | 13 | 23
  1-3 years | 14 | 9 | 23
  Greater than 3 years | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Patient Numerical Pain Ranking Scale (NPRS)
Description: Validated pain scale, subject reported. Min 0, Max 10, Higher score means worse outcome.
Time Frame: 6 weeks after surgery date
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
score on a scale | 1.8 [1.3 to 2.3] | 2.3 [1.7 to 2.9]

2. Secondary Outcome: HOOS - Hip Disability and Osteoarthritis Outcome Score
Description: questionnaire used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process. Min 0, Max 100. Lower score means worse outcome.
Time Frame: at 6 week and 6 month after surgery date
Population: There was patient drop out between 6 week and 6 month time points, which is why there are fewer patients at the 6 month time point.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
score on a scale
  6 week | 73.9 [68.5 to 79.3] | 71.6 [65.9 to 77.3]
  6 month: number analyzed (Participants) | 30 | 27
  6 month | 83.4 [77.7 to 89.1] | 80.8 [74.0 to 87.7]

3. Secondary Outcome: VR12 - Veteran RAND 12 Item Health Survey
Description: general health outcome survey. The results of the VR-12 are summarized as two scores - a Mental Component Score (MCS) and a Physical Component Score (PCS). The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). The United States population average PCS and MCS are both 50 points. The United States population standard deviation is 10 points. Therefore, each increment of 10 points above or below 50 corresponds to one standard deviation away from the population average.
Time Frame: at 6 week and 6 month after surgery date
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
score on a scale
  Mental Component Summary 6 weeks | 53.1 [50.2 to 56.1] | 49.0 [44.8 to 53.3]
  Physical Component Summary 6 weeks | 38.2 [34.4 to 42.0] | 37.1 [33.7 to 40.6]
  Mental Component Summary 6 months: number analyzed (Participants) | 30 | 27
  Mental Component Summary 6 months | 52.2 [48.1 to 56.3] | 51.1 [46.9 to 55.3]
  Physical Component Summary 6 months: number analyzed (Participants) | 30 | 27
  Physical Component Summary 6 months | 47.0 [43.6 to 50.4] | 46.3 [42.6 to 50.0]

4. Secondary Outcome: Patient Using Topical Non-steroidal Medication
Description: Number of patient using a topical nonsteroidal medication is listed here.
Time Frame: 6 week and 6 month after surgery date
Population: There was patient drop out between 6 week and 6 month time points, which is why there are fewer patients at the 6 month time point. Additionally, at the 6 month mark we have HOOS outcome scores for a higher number of patients than we have this secondary outcome measures due to incomplete final capture of information at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
Participants
  6 week | 1 | 3
  6 month: number analyzed (Participants) | 28 | 25
  6 month | 1 | 2

5. Secondary Outcome: Patient Received Cortisone Injection to Hip Flexor Sheath or Bursa
Description: Number of patients who received a cortisone injection to hip flexor sheath or bursa is listed here.
Time Frame: 6 week and 6 month after surgery date
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
Participants
  6 week | 0 | 0
  6 month: number analyzed (Participants) | 28 | 25
  6 month | 4 | 0

6. Secondary Outcome: Patient Using Opioid Medication
Description: Number of patients using opioids is listed here.
Time Frame: 6 week and 6 month after surgery date
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 37 | 36
Participants
  6 week | 2 | 1
  6 month: number analyzed (Participants) | 28 | 25
  6 month | 1 | 0

7. Secondary Outcome: NPRS - Numerical Pain Ranking Scale
Description: Validated pain scale, subject reported. Min 0, Max 10, Higher score means worse outcome.
Time Frame: 6 months after surgery date
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Hip Brace | No Brace
Number analyzed (Participants) | 30 | 27
score on a scale | 1.6 [1.0 to 2.3] | 1.9 [1.1 to 2.6]

ADVERSE EVENTS:
Time Frame: 6 months for each patient
Description: No difference from set definitions.
Arm/Group | Hip Brace | No Brace
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/36
Other Adverse Events (participants affected / at risk) | 3/37 | 2/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hip Brace (N=37) | No Brace (N=36)
Numbness (Nervous system disorders) | 3 (3) | 2 (2) — Temporary decrease sensation on operative extremity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04599296/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT04599296/ICF_001.pdf